CLINICAL TRIAL: NCT03351244
Title: A Phase II Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Orally Administered BI 409306 During a 28-week Treatment Period as Adjunctive Therapy to Antipsychotic Treatment for the Prevention of Relapse in Patients With Schizophrenia.
Brief Title: This Study Tests Whether BI 409306 Prevents Patients With Schizophrenia From Becoming Worse. This Study Looks at How Well Patients Tolerate BI 409306 and How Effective it is Over 6 Months
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: disruption due to COVID-19
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1289-0049; 2017-002369-23 (EudraCT Number)
Record Dates: First submitted 2017-11-20; First posted 2017-11-22 (Actual); Results first posted 2022-04-04 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — BI 409306

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BI 409306 50 mg (Experimental): 1 film-coated tablet of 50 milligrams (mg) of BI 409306 plus 1 tablet of 25 mg matching placebo were administered orally once daily for a treatment period of 28 weeks, followed by a withdrawal/taper period of 7 days, followed by a follow-up period of 3 weeks.
  Interventions: Drug: BI 409306
- BI 409306 25 mg (Experimental): 1 film-coated tablet of 25 milligrams (mg) of BI 409306 plus 1 tablet of 50 mg matching placebo were administered orally once daily for a treatment period of 28 weeks, followed by a withdrawal/taper period of 7 days, followed by a follow-up period of 3 weeks.
  Interventions: Drug: BI 409306
- Placebo (Placebo Comparator): 1 film-coated tablet of 25 milligrams (mg) of matching Placebo plus 1 tablet of 50 mg matching placebo were administered orally once daily for a treatment period of 28 weeks, followed by a withdrawal/taper period of 7 days, followed by a follow-up period of 3 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 409306 — 28 week treatment period
  Arms: BI 409306 25 mg; BI 409306 50 mg
Drug: Placebo — 28 week treatment period
  Arms: Placebo

SUMMARY:
The objective of the study is to investigate the efficacy, safety and tolerability of BI 409306 once daily compared with placebo given for 28 weeks in patients with schizophrenia on antipsychotic treatment. The study is designed to show superiority of BI 409306 over placebo in preventing relapse of schizophrenia symptoms.

ELIGIBILITY:
Inclusion Criteria:

* International Statistical Classification of Diseases and Related Health Problems, 10th Revision (ICD-10) diagnosis of schizophrenia >= one year prior to randomisation.
* Outpatients in the stable phase of illness, as assessed by the investigator after review of medical records or documented discussion with treating clinician.
* Patients currently taking a stable dose of antipsychotic medication(s) for at least 12 weeks prior to randomisation.
* Detectable level of current antipsychotic medication(s) in plasma from blood drawn at Visit 1 (unless no assay is available for the antipsychotic(s) currently prescribed).
* Patients who have experienced at least 2 relapses within the past 5 years or at least 1 relapse if they were diagnosed less than 3 years ago. Relapse is defined as the patient having any of the following using the above number of relapses and time frames:

  * Hospitalization for psychosis (involuntary or voluntary admission), intensive outpatient therapy or use of home treatment as an alternative to hospitalization (verified via medical record).
  * Emergency Department visit for worsening schizophrenia symptoms (verified via medical record).
  * Deliberate self-injury and/or violent behaviour resulting in significant injury to another person or property (verified by police record or treating mental health provider written record or documented phone conversation).
  * Change in the patient's antipsychotic medication or increase in antipsychotic medication dosage due to worsening of schizophrenia symptoms (verified by pharmacy records or treating mental health provider written record or documented phone conversation).
* Clinical Global Impressions-Severity (CGI-S) score ≤4 at Visit 1 and 2.
* Positive and Negative Syndrome Scale (PANSS) total score <80 and a score of ≤ 4 on individual PANSS items conceptual disorganization, hallucinatory behavior, suspiciousness, and unusual thought content at Visit 1.
* Of full age (according to local legislation, usually ≥ 18 years) and ≤ 55 years at the time of informed consent.
* Patients must have an identified informant who will be consistent throughout the study.
* Patients who report living at the same address for the 3 months prior to randomisation.
* Male or female patients.

  -- Female patients of childbearing potential must be ready and able to use highly effective methods of birth control per International Conference on Harmonisation (ICH) M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. Patients must agree to use birth control throughout the trial and for at least 28 days after treatment has ended. Acceptable methods of birth control include combined estrogen-progestin oral, intravaginal or transdermal contraceptives, progestogen-only oral, injectable or implantable contraceptives, intrauterine devices (IUDs), intrauterine hormone releasing systems (IUSs), bilateral tubal occlusion, vasectomized sexual partner, and complete sexual abstinence (if acceptable by local health authorities) is allowed when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptom-thermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Male patients who are able to father a child must be ready and able to be abstinent or use adequate contraception for the duration of study participation and for at least 28 days after treatment has ended.
* Signed and dated written informed consent in accordance with International Conference on Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial. If the patient has a legal representative, then this legal representative must give written informed consent as well.

Exclusion criteria:

* Patients treated with more than two antipsychotic medications (including more than two dosage forms).
* Patients who are currently being treated with clozapine, or who have been treated with clozapine in the past 5 years.
* Patients with a categorical diagnosis of another current major psychiatric disorder per the Mini-international neuropsychiatric Interview (M.I.N.I.).
* Homicidal behaviour (in the investigator's judgement) in the past 2 years.
* Any suicidal behavior in the past 2 years (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior).
* Any suicidal ideation of type 4 or 5 in the Columbia Suicide Severity Rating Scale (CSSRS) in the past 3 months (i.e. active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent).
* In the judgment of the investigator, any clinically significant finding from the physical examination or laboratory value deviating from normal or any evidence of a clinically significant concomitant disease or any other clinical condition that would jeopardize a patient's safety while participating in the clinical trial.
* Other known neurological diseases (including but not limited to any kind of seizures or stroke).
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix.
* Planned elective surgery requiring general anesthesia, or hospitalization for more than 1 day during the study period.
* Significant history of drug or alcohol dependence or abuse (Substance Use Disorder as defined in Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) or ICD-10) within the last six months prior to informed consent. (Not including caffeine or nicotine).
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
* Patients taking strong or moderate CYP1A2 inhibitors who are also a CYP2C19 Poor Metabolizer (PM). Patients taking medication known to be strong or moderate inhibitors of CYP1A2 must be prospectively genotyped to ensure they are not poor metabolizers of CYP2C19. (A list of CYP1A2 and CYP2C19 inhibitors can be found in the Investigator Site File (ISF)).
* Patients taking strong or moderate CYP1A2 inhibitors who are also taking concomitant strong or moderate CYP2C19 inhibitors. (A list of CYP1A2 and CYP2C19 inhibitors can be found in the ISF)
* Patients with a history of moderate to severe hepatic impairment (Child-Pugh B / C).
* Patients with a history of moderate to severe renal impairment (Stage 3 - 5).
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
* In the judgment of the investigator, inability of the patient to comply with the clinical trial procedures.
* Currently enrolled in another investigational device or drug study, or less than 6 months from Visit 1 since ending another investigational device or drug study(s), or participation in > 2 investigational drug clinical trials in the past 2 years.
* Previous randomisation in any BI 409306 study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 264 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (59):
- United States (32):
  - Alea Research, Phoenix, Arizona
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Collaborative Neuroscience Network, LLC (CNS), Garden Grove, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Synergy East, Lemon Grove, California
  - University of California Los Angeles, Los Angeles, California
  - Excell Research Inc., Oceanside, California
  - Orange County Neuropsychiatric Research Center LLC, Orange, California
  - Collaborative Neuroscience Network, LLC (CNS), Torrance, California
  - MD Clinical, Hallandale, Florida
  - Reliable Clinical Research, Hialeah, Florida
  - Meridien Research, Maitland, Florida
  - Behavioral Clinical Research, Inc., North Miami, Florida
  - Meridien Research, Orlando, Florida
  - Atlanta Center, Atlanta, Georgia
  - Alam Medical Research, Inc., Chicago, Illinois
  - Lake Charles Clinical Trials LLC, Lake Charles, Louisiana
  - Clinical Trials of America, LLC, Monroe, Louisiana
  - Michigan Clinical Research Institute PC, Ann Arbor, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - St. Charles Psychiatric Associates & Midwest Research Group, Saint Charles, Missouri
  - Arch Clinical Trials, St Louis, Missouri
  - PsychCare Consultants Research, St Louis, Missouri
  - Altea Research Institute, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - New York State Psychiatric Institute, New York, New York
  - Manhattan Behavioral Medicine PLLC, New York, New York
  - Community Clinical Research, Inc., Austin, Texas
  - University Hills Clinical Research, Irving, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas
  - @Health Texas, Richmond, Texas
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - Dr. Alexander McIntyre Inc., Penticton, British Columbia
  - The Medical Arts Health Research Group, Vancouver, British Columbia
  - Chatham-Kent Clinical Trials Research Centre, Chatham, Ontario
  - Centre for Addiction and Mental Health (CAMH), Toronto, Ontario
  - IUSMM Institut Universitaire en Sante Mentale de Montreal, Montreal, Quebec
- France (5):
  - HOP la Colombière, Montpellier
  - GHU Paris Psychiatrie et Neurosciences, Paris
  - HOP Guillaume Régnier, Rennes
  - HOP Nord, Saint-Priest-en-Jarez
  - HOP Sainte Musse, Toulon
- Japan (10):
  - Okehazama Hospital Fujita Kokoro Care Center, Aichi, Toyoake
  - Fujita Health University Hospital, Aichi, Toyoake
  - National Center for Global Health and Medicine Kohnodai Hospital, Chiba, Ichikawa
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Kuramitsu Hospital, Fukuoka, Fukuoka
  - Soushu Hospital, Kanagawa, Atsugi
  - Kishiro Mental Clinic, Kanagawa, Kawasaki
  - Nara Medical University Hospital, Nara, Kashihara
  - National Hospital Organization Hizen Psychiatric Medical Center, Saga, Kanzaki-gun
  - National Center Neurology and Psychiatry, Tokyo, Kodaira
- South Korea (3):
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
- Hospital Universitario Marqués de Valdecilla, Santander, Spain
- Taiwan (2):
  - NCKUH, Tainan
  - Taoyuan Psychiatric Center, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a "Document Sharing Agreement". For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Zhu Z, Roy D, Feng S, Vogler B. AI-based medication adherence prediction in patients with schizophrenia and attenuated psychotic disorders. Schizophr Res. 2025 Jan;275:42-51. doi: 10.1016/j.schres.2024.11.006. Epub 2024 Dec 4. PMID 39637767
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase II trial aimed to evaluate the impact of 28-week treatment with BI 409306 (added to standard antipsychotic medication) compared with placebo on preventing relapse in patients with schizophrenia.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 409306 25 mg: 1 film-coated tablet of 25 milligrams (mg) of BI 409306 plus 1 tablet of 50 mg matching placebo were administered orally once daily for a treatment period of 28 weeks, followed by a withdrawal/taper period of 7 days, followed by a follow-up period of 3 weeks.
  Participants were randomized to either withdrawal or taper period in 1:1 ratio at the randomization of treatment groups.
  Withdrawal period: 4 tablets of 10 mg placebo once daily (q.d.) on Day 1 of withdrawal period; 3 tablets of 10 mg placebo q.d. on Day2-3 of withdrawal period; 2 tablets of 10mg placebo q.d. on Day 4-5 of withdrawal period; 1 tablet of 10mg placebo q.d. on Day 6-7 of withdrawal period.
  Taper period: 2 tablets of 10 mg BI 409306 and 2 tablets of placebo q.d. on Day 1 of the taper period; 2 tablets of 10 mg BI 409306 and 1 tablet of placebo q.d. on Day 2-3 of taper period; 1 tablet of 10 mg BI 409306 and 1 tablet of placebo q.d. on Day 4-5 of taper period; 1 tablet of 10 mg BI 409306 q.d. on Day 6-7 of taper period.
- BI 409306 50 mg: 1 film-coated tablet of 50 milligrams (mg) of BI 409306 plus 1 tablet of 25 mg matching placebo were administered orally once daily for a treatment period of 28 weeks, followed by a withdrawal/taper period of 7 days, followed by a follow-up period of 3 weeks.
  Participants were randomized to either withdrawal or taper period in 1:1 ratio at the randomization of treatment groups.
  Withdrawal period: 4 tablets of 10 mg placebo once daily (q.d.) on Day 1 of withdrawal period; 3 tablets of 10 mg placebo q.d. on Day2-3 of withdrawal period; 2 tablets of 10mg placebo q.d. on Day 4-5 of withdrawal period; 1 tablet of 10mg placebo q.d. on Day 6-7 of withdrawal period.
  Taper period: 4 tablets of 10 mg BI 409306 q.d. on Day 1 of taper period; 3 tablets of 10 mg BI 409306 q.d. on Day 2-3 of taper period; 2 tablets of 10 mg BI 409306 q.d. on Day 4-5 of taper period; 1 tablet of 10 mg BI 409306 q.d. on Day 6-7 of taper period.
- Placebo: 1 film-coated tablet of 25 milligrams (mg) of matching Placebo plus 1 tablet of 50 mg matching placebo were administered orally once daily for a treatment period of 28 weeks, followed by a withdrawal/taper period of 7 days, followed by a follow-up period of 3 weeks.
  Participants were randomized to either withdrawal or taper period in 1:1 ratio at the randomization of treatment groups.
  Both withdrawal and taper periods: 4 tablets of 10 mg placebo once daily (q.d.) on Day 1 of withdrawal/taper period; 3 tablets of 10 mg placebo q.d. on Day 2-3 of withdrawal/taper period; 2 tablets of 10mg placebo q.d. on Day 4-5 of withdrawal/taper period; 1 tablet of 10mg placebo q.d. on Day 6-7 of withdrawal/taper period.
Period: Overall Study
Arm/Group | BI 409306 25 mg | BI 409306 50 mg | Placebo
Started | 89 | 88 | 87
Completed | 62 | 48 | 53
Not Completed | 27 | 40 | 34
Not completed — Adverse Event | 7 | 11 | 12
Not completed — Investigator's decision | 0 | 0 | 2
Not completed — System error | 0 | 0 | 2
Not completed — COVID-19 restrictions | 3 | 0 | 1
Not completed — Non-compliance | 2 | 5 | 0
Not completed — Withdrawal by Subject | 11 | 16 | 13
Not completed — Lost to Follow-up | 2 | 6 | 4
Not completed — Protocol Violation | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): the TS includes all patients who were randomised and were documented to have taken at least 1 dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 409306 25 mg | BI 409306 50 mg | Placebo | Total
Number analyzed (Participants) | 89 | 88 | 87 | 264
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.4 (9.8) | 41.9 (9.6) | 40.5 (9.8) | 40.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 36 | 32 | 97
  Male | 60 | 52 | 55 | 167
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 15 | 15 | 40
  Not Hispanic or Latino | 75 | 69 | 68 | 212
  Unknown or Not Reported | 4 | 4 | 4 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 23 | 20 | 20 | 63
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  Black or African American | 36 | 37 | 32 | 105
  White | 23 | 24 | 25 | 72
  More than one race | 1 | 1 | 2 | 4
  Unknown or Not Reported | 6 | 4 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of First Relapse After 28 Weeks of Treatment
Description: The incidence rate of first relapse after 28 weeks of treatment is reported. For each treatment group, the incidence rate was calculated as the number of events / sum of the observational time (patient year) over all participants in this treatment group.
Time Frame: 28 weeks
Population: Full analysis set (FAS): the FAS includes all patients in the treated set with at least 1 baseline and post-baseline measurement of any type.
Measure: Number; unit: Events per patient-years
Groups:
- BI 409306 Pooled: This group included all participants who administered BI 409306 during the study.
Arm/Group | BI 409306 25 mg | BI 409306 50 mg | BI 409306 Pooled | Placebo
Number analyzed (Participants) | 89 | 88 | 177 | 87
Events per patient-years | 0.527 | 0.434 | 0.482 | 0.496
Statistical Analysis 1: Comparison: BI 409306 25 mg vs Placebo; Test type: Other; p = 0.7735, Regression, Cox; The model included the treatment effect as the only covariate and was stratified by country; Hazard Ratio (HR) = 1.097, 95% CI 2-sided [0.585 to 2.056]
Statistical Analysis 2: Comparison: BI 409306 50 mg vs Placebo; Test type: Other; p = 0.7809, Regression, Cox; The model included the treatment effect as the only covariate and was stratified by country; Hazard Ratio (HR) = 0.910, 95% CI 2-sided [0.468 to 1.770]
Statistical Analysis 3: Comparison: BI 409306 Pooled vs Placebo; Test type: Other; p = 0.9862, Regression, Cox; The model included the treatment effect as the only covariate and was stratified by country; Hazard Ratio (HR) = 1.005, 95% CI 2-sided [0.576 to 1.753]

2. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Positive Symptoms Score After 28 Weeks of Treatment
Description: Positive and Negative Syndrome Scale (PANSS): assesses the severity of psychotic symptoms and progression of disease.
  The PANSS positive symptoms score is the sum of scores from 7 Items where each item has a minimum score 1 (better outcome) and maximum score 7 (worse outcome). The PANSS positive symptoms score ranges from 7 (less severe the disease) to 49 (more severe the disease).
Time Frame: At baseline and at Week 28.
Population: Full analysis set (FAS): the FAS includes all patients in the treated set with at least 1 baseline and post-baseline measurement of any type. Only participants with non-missing results were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | BI 409306 25 mg | BI 409306 50 mg | BI 409306 Pooled | Placebo
Number analyzed (Participants) | 73 | 55 | 128 | 65
Score on a scale | -0.54 [-1.370 to 0.294] | -0.71 [-1.641 to 0.224] | -0.61 [-1.231 to 0.005] | -0.92 [-1.769 to -0.070]
Statistical Analysis 1: Comparison: BI 409306 25 mg vs Placebo; Test type: Other — A restricted maximum likelihood-based approach using a mixed model with repeated measurements was applied; p = 0.5289, Mixed model with repeated measurements; The analysis included the fixed, categorical effects of treatment at each visit, and the fixed continuous effects of baseline at each visit; Placebo-corrected adjusted mean = 0.38, 95% CI 2-sided [-0.809 to 1.570]
Statistical Analysis 2: Comparison: BI 409306 50 mg vs Placebo; Test type: Other — A restricted maximum likelihood-based approach using a mixed model with repeated measurements was applied; p = 0.7440, Mixed model with repeated measurements; [statistical method as in outcome 2, analysis 1]; Placebo-corrected adjusted mean = 0.21, 95% CI 2-sided [-1.055 to 1.475]
Statistical Analysis 3: Comparison: BI 409306 Pooled vs Placebo; Test type: Other — A restricted maximum likelihood-based approach using a mixed model with repeated measurements was applied; p = 0.5659, Mixed model with repeated measurements; [statistical method as in outcome 2, analysis 1]; Placebo-corrected adjusted mean = 0.31, 95% CI 2-sided [-0.745 to 1.358]

3. Secondary Outcome: Change From Baseline in Clinical Global Impressions-Severity (CGI-S) Scale Score After 28 Weeks of Treatment
Description: Clinical Global Impressions-Severity (CGI-S): One-item evaluation completed by the clinician to measure the severity of psychopathology.
  The CGI-S score ranges from 1 (normal) through to 7 (most severely ill). The higher the score, the worse the psychopathology.
Time Frame: At baseline and at Week 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BI 409306 25 mg | BI 409306 50 mg | BI 409306 Pooled | Placebo
Number analyzed (Participants) | 73 | 55 | 128 | 65
Score on a scale | -0.15 (0.758) | -0.22 (0.839) | -0.18 (0.791) | -0.22 (0.718)

4. Secondary Outcome: Patient Global Impressions-Improvement (PGI-I) Scale Score After 28 Weeks of Treatment
Description: Patient Global Impressions-Improvement (PGI-I): One-item evaluation completed by the patient to assess their overall evaluation of his/her status compared to how they felt at randomisation.
  The PGI-I score ranges from 1 (Very much better) through to 7 (Very much worse). The higher the score, the worse the improvement.
Time Frame: At Week 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BI 409306 25 mg | BI 409306 50 mg | BI 409306 Pooled | Placebo
Number analyzed (Participants) | 72 | 54 | 126 | 63
Score on a scale | 2.61 (1.328) | 2.96 (1.197) | 2.76 (1.280) | 2.94 (1.190)

5. Secondary Outcome: Incidence Rate of Suicidal Ideation and Behaviour (Assessed by Columbia Suicide Severity Rating Scale (C-SSRS)) After 28 Weeks of Treatment
Description: Columbia Suicide Severity Rating Scale (C-SSRS): suicide risk assessment. At a minimum, the interview consists of 2 screening questions related to suicidal ideation and 4 related to suicidal behavior, and may be expanded to up to 17 items in case of positive responses. Free text entries are allowed.
  Suicidal behavior is collected in nominal scale as presence/absence of actual attempts, non-suicidal self-injurious behavior, interrupted attempts, aborted attempts, preparatory acts or behavior, and any suicidal behavior.
  Suicidal ideation is rated on a 6-point scale from 0 (No ideation present) to 5 (Active ideation with plan and intent). A score of 4 or 5 on this scale indicates serious suicidal ideation.
  For each treatment group, the incidence rate was calculated as the number of events / sum of the observational time (patient year) over all participants in this treatment group.
Time Frame: 28 weeks
Population: as for outcome 1
Measure: Number; unit: Events per patient-years
Arm/Group | BI 409306 25 mg | BI 409306 50 mg | BI 409306 Pooled | Placebo
Number analyzed (Participants) | 89 | 88 | 177 | 87
Events per patient-years | 0.070 | 0.077 | 0.073 | 0.071
Statistical Analysis 1: Comparison: BI 409306 25 mg vs Placebo; Test type: Other; p = 0.9938, Regression, Cox; The model included the treatment effect as the only covariate and was stratified by country; Hazard Ratio (HR) = 1.006, 95% CI 2-sided [0.203 to 4.989]
Statistical Analysis 2: Comparison: BI 409306 50 mg vs Placebo; Test type: Other; p = 0.8930, Regression, Cox; The model included the treatment effect as the only covariate and was stratified by country; Hazard Ratio (HR) = 1.116, 95% CI 2-sided [0.225 to 5.531]
Statistical Analysis 3: Comparison: BI 409306 Pooled vs Placebo; Test type: Other; p = 0.9360, Regression, Cox; The model included the treatment effect as the only covariate and was stratified by country; Hazard Ratio (HR) = 1.058, 95% CI 2-sided [0.265 to 4.233]

6. Secondary Outcome: Change From Baseline in Personal and Social Performance Scale (PSP) Score After 28 Weeks of Treatment
Description: Personal and Social Performance scale (PSP): The PSP is a 100-point, single item, clinician rated scale to assess 4 domains of social functioning (Four domains over the past month: (1) socially useful activities, (2) personal and social relationships, (3) self-care and (4) disturbing and aggressive behaviors.) in patients with schizophrenia. The PSP score is a single score ranging from 1 to 100. Higher scores represent better personal and social functioning.
Time Frame: At baseline and at Week 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BI 409306 25 mg | BI 409306 50 mg | BI 409306 Pooled | Placebo
Number analyzed (Participants) | 72 | 54 | 126 | 65
Score on a scale | 2.8 (8.8) | 2.4 (9.4) | 2.6 (9.1) | 3.0 (10.2)

7. Secondary Outcome: Incidence Rate of New Prescription or Increase in Dose of an Ongoing Antipsychotic Medication
Description: The incidence rate of new prescription or increase in dose of an ongoing antipsychotic medication is reported. For each treatment group, the incidence rate was calculated as the number of events / sum of the observational time (patient year) over all participants in this treatment group.
Time Frame: 28 weeks
Population: as for outcome 1
Measure: Number; unit: Events per patient-years
Arm/Group | BI 409306 25 mg | BI 409306 50 mg | BI 409306 Pooled | Placebo
Number analyzed (Participants) | 89 | 88 | 177 | 87
Events per patient-years | 0.168 | 0.130 | 0.149 | 0.217
Statistical Analysis 1: Comparison: BI 409306 25 mg vs Placebo; Test type: Other; p = 0.6362, Regression, Cox; The model included the treatment effect as the only covariate and was stratified by country; Hazard Ratio (HR) = 0.788, 95% CI 2-sided [0.293 to 2.118]
Statistical Analysis 2: Comparison: BI 409306 50 mg vs Placebo; Test type: Other; p = 0.3782, Regression, Cox; The model included the treatment effect as the only covariate and was stratified by country; Hazard Ratio (HR) = 0.612, 95% CI 2-sided [0.205 to 1.826]
Statistical Analysis 3: Comparison: BI 409306 Pooled vs Placebo; Test type: Other; p = 0.4253, Regression, Cox; The model included the treatment effect as the only covariate and was stratified by country; Hazard Ratio (HR) = 0.703, 95% CI 2-sided [0.296 to 1.671]

ADVERSE EVENTS:
Time Frame: All-cause mortality: From first dose until withdraw or end of 1-week taper period + 3-week follow-up period, up to 32 weeks. Serious (non-serious) adverse events: From first dose until withdraw or end of 1-week taper period + 1-week residual effect period, up to 30 weeks.
Description: Treated set (TS): the TS includes all patients who were randomised and were documented to have taken at least 1 dose of trial drug.
Groups:
- Total: All participants randomised in this study.
Arm/Group | BI 409306 25 mg | BI 409306 50 mg | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/89 | 1/88 | 0/87 | 1/264
Serious Adverse Events (participants affected / at risk) | 9/89 | 7/88 | 12/87 | 28/264
Other Adverse Events (participants affected / at risk) | 30/89 | 25/88 | 19/87 | 74/264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 409306 25 mg (N=89) | BI 409306 50 mg (N=88) | Placebo (N=87) | Total (N=264)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Complicated appendicitis (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 3 | 3
Wound infection (Infections and infestations) | 0 | 0 | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Acute psychosis (Psychiatric disorders) | 1 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1
Delusion (Psychiatric disorders) | 0 | 0 | 1 | 1
Depression suicidal (Psychiatric disorders) | 0 | 0 | 1 | 1
Hallucination, auditory (Psychiatric disorders) | 1 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 1 | 0 | 2
Schizophrenia (Psychiatric disorders) | 2 | 1 | 4 | 7
Substance abuse (Psychiatric disorders) | 1 | 0 | 0 | 1
Suicidal behaviour (Psychiatric disorders) | 0 | 1 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 3 | 0 | 2 | 5
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 409306 25 mg (N=89) | BI 409306 50 mg (N=88) | Placebo (N=87) | Total (N=264)
Photophobia (Eye disorders) | 3 | 8 | 1 | 12
Vomiting (Gastrointestinal disorders) | 1 | 1 | 5 | 7
Nasopharyngitis (Infections and infestations) | 7 | 5 | 7 | 19
Headache (Nervous system disorders) | 6 | 7 | 4 | 17
Somnolence (Nervous system disorders) | 5 | 3 | 3 | 11
Insomnia (Psychiatric disorders) | 5 | 6 | 0 | 11
Schizophrenia (Psychiatric disorders) | 6 | 4 | 2 | 12

LIMITATIONS AND CAVEATS:
The study was terminated due to sponsor decision. The planned number of participants to be recruited was not reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT03351244/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT03351244/SAP_001.pdf